CLINICAL TRIAL: NCT04639011
Title: Effects of Duloxetine on Postoperative Pain Control and Knee Rehabilitation After Open Reduction Internal Fixation of Tibial Plateau Fractures
Brief Title: Duloxetine Tibial Plateau
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not conducted because funding was not obtained.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-40569
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Tibial Plateau Fracture; Pain, Postoperative
Keywords: Duloxetine; VAS pain scores; Patient Controlled Analgesia (PCA)
MeSH Terms: conditions — Tibial Plateau Fractures; Pain, Postoperative | interventions — Duloxetine Hydrochloride; Sugars; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A Placebo (Active Comparator): Participants randomized to Group A will receive placebo (sugar pill) and Boston Medical Center (BMC) standard of care.
  Interventions: Other: Placebo; Other: Standard of care (SOC) for tibial plateau surgery
- Groups B Intervention (Experimental): Participants randomized to Group B will receive duloxetine and Boston Medical Center (BMC) standard of care.
  Interventions: Drug: Duloxetine; Other: Standard of care (SOC) for tibial plateau surgery

INTERVENTIONS:
Drug: Duloxetine — Three doses of 60 mg of oral duloxetine will be given to participants (right before operation, postop day 1, postop day 2)
  Other Names: Serotonin-norepinephrine reuptake inhibitor (SNRI)
  Arms: Groups B Intervention
Other: Placebo — Three doses of placebo will be given to participants (right before operation, postop day 1, postop day 2).
  Other Names: Sugar pill
  Arms: Group A Placebo
Other: Standard of care (SOC) for tibial plateau surgery — Postoperative IV administration of opioids via a patient controlled analgesia (PCA) system which utilizes a hydromorphone pump.

SUMMARY:
The purpose of this study is to determine if Duloxetine provides effective pain management for adult patients (18 or older) undergoing tibial plateau surgery. Participants from two institutions will be randomized to one of two treatment groups: control (Group A) and treatment (Group B). Group A control group will receive placebo of sugar pill and BMC standard of care - namely postoperative, IV administration of opioids via a patient controlled analgesia (PCA) system which utilizes a hydromorphone pump (BMC standard of care). Group B, the intervention group, will receive three doses of 60 mg of oral duloxetine (right before operation, postop day 1, postop day 2).

This study is important as tibial plateau surgery's postoperative pain management primarily involved providing opioids, and if duloxetine can result in reduced narcotic intake and lower pain scores, it can potentially improve patient care, rehabilitation, early movement, and shorter length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Tibial plateau fracture that requires operative fixation
* Ambulatory patient prior to fracture

Exclusion Criteria:

* Previous tibial plateau fracture on ipsilateral knee
* History of Complex Regional Pain Syndrome in ipsilateral extremity
* History of any demyelinating disorder or neurologic deficit that may contribute to altered pain tolerance/sensation
* Acute or chronic knee infection in ipsilateral extremity
* Previous total knee arthroplasty or knee hemiarthroplasty in ipsilateral knee
* Allergy to morphine (used in the SOC PCA pump)
* Pregnant or breastfeeding as determined by standard of care pre-operative urine pregnancy test
* Polytrauma
* Open fracture
* IV drug user
* Rheumatoid arthritis
* Revision cases
* Non-ambulatory
* Anatomical deformities of the knee
* Hepatic dysfunction or cirrhosis
* Taking Selective Serotonin Reuptake Inhibitor (SSRI), serotonin-norepinephrine reuptake Inhibitor (SNRI), monoamine oxidase inhibitors (MAOIs), tri- or tetra- cyclic anti-depressant
* Renal impairment (mention in patient chart and/or creatinine clearance <30)
* Moderate to severe depression
* Taking CYP1A2 inhibitors and CYP1A6 inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain levels in the first 16 hours after surgery | every 4 hours up to 16 hours
  A visual analog pain scale (VAS) will be used to assess postoperative pain levels. Participants will make a mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." HIgher scores reflect greater pain levels.
Pain level 24 hours after surgery | 24 hours
  A visual analog pain scale (VAS) will be used to assess the postoperative pain level. Participants will make a mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." HIgher scores reflect greater pain levels.
Pain level 36 hours after surgery | 36 hours
  A visual analog pain scale (VAS) will be used to assess the postoperative pain level. Participants will make a mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." HIgher scores reflect greater pain levels.

SECONDARY OUTCOMES:
Total morphine consumption | up to 10 days post op
  The total morphine consumption will be calculated using the Centers for Disease Control (CDC) morphine equivalents [ME].Determine the total daily amount of morphine taken; convert to MEs by multiplying the daily dosage for each opioid by its conversion factor [which is =1 for morphine]; then add all morphine MEs together.
Change in knee range of motion | 6 weeks, 12 weeks
  The knee range of motion will be abstracted from the electronic medical record. Knee range of motion ranges from 0 to 140 degrees.
Self reported functional status at 6 weeks | 6 weeks
  Functional status will be assessed using the Short Musculoskeletal Function Assessment (SMFA). SMFA is a 46 item questionnaire. It consists of the dysfunction index, which has 34 items for the assessment of patient function, and the bother index, which has 12 items for the assessment of how much patients are bothered by functional problems.
Self reported functional status at 12 weeks | 12 weeks
  Functional status will be assessed using the Short Musculoskeletal Function Assessment (SMFA). SMFA is a 46 item questionnaire. It consists of the dysfunction index, which has 34 items for the assessment of patient function, and the bother index, which has 12 items for the assessment of how much patients are bothered by functional problems.
Hospital length of stay | 12 weeks
  The hospital length of stay will be measured in days, calculated by subtracting the date of admission from the date of discharge as recorded in the electronic medical record.
Time to mobilization (starting to walk) | 12 weeks
  The time to mobilization will be calculated by subtracting the date the participant started to walk post operatively from the date of surgery as recorded in the electronic medical record.
Ambulation (walking) distance on post-op days 1 or 2 | Up to 2 days post op
  The walking distance will be abstracted from the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Seroos Salavati, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Westchester Medical Center, Valhalla, New York

IPD SHARING:
Plan to Share IPD: No